CLINICAL TRIAL: NCT04222595
Title: FluPRINT Study OVG 2018/04: Characterisation of the Immune & Transcriptional Responses to Live Attenuated Influenza Vaccine (LAIV) in Healthy 4-6-year-old Children
Brief Title: FluPRINT Study: Characterisation of the Immune and Transcriptional Response to LAIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European Commission (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FluPRINT Study OVG 2018/04
Record Dates: First submitted 2018-10-17; First posted 2020-01-10 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2021-01

CONDITIONS: Immunization
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Open-label study of healthy and immunocompetent children aged 4 to 6 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1- naive (No Intervention): Group 1: up to 10 children aged 4-6 years that never received LAIV before.
- 2- Fluenz Tetra nasal spray suspension (Active Comparator): Group 2: up to 10 children aged 4-6 years that received LAIV once before. Single dose vaccine, administered as a nasal spray (0.2 ml administered as 0.1 ml per nostril).
  Interventions: Other: Fluenz Tetra nasal spray suspension
- 3- Fluenz Tetra nasal spray suspension (Active Comparator): Group 3: up to 10 children aged 4-6 years that were vaccinated twice before.Single dose vaccine, administered as a nasal spray (0.2 ml administered as 0.1 ml per nostril).
  Interventions: Other: Fluenz Tetra nasal spray suspension
- 4- Fluenz Tetra nasal spray suspension (Active Comparator): Group 4: up to 10 children aged 4-6 years that were vaccinated 3 or 4 times before.Single dose vaccine, administered as a nasal spray (0.2 ml administered as 0.1 ml per nostril).
  Interventions: Other: Fluenz Tetra nasal spray suspension

INTERVENTIONS:
Other: Fluenz Tetra nasal spray suspension — Prophylaxis of influenza in children and adolescents from 24 months to less than 18 years of age. Single dose vaccine, administered as a nasal spray (0.2 ml administered as 0.1 ml per nostril).
  Other Names: Influenza vaccine (live attenuated, nasal)
  Arms: 2- Fluenz Tetra nasal spray suspension; 3- Fluenz Tetra nasal spray suspension; 4- Fluenz Tetra nasal spray suspension

SUMMARY:
In 2013 the UK government introduced the nasal flu spray vaccine (Fluenz Tetra®) for use in children from 24 months to less than 18 years of age. This is a licensed vaccine that is safe, effective and like the injectable vaccine, needs to be given yearly. There is evidence that the nasal spray flu vaccine can offer better protection for children than the injectable flu vaccine but it is not yet fully understood why this is so. When the immune system responds to an infection or a vaccine, specific 'immune response' genes are activated or 'switched on'. This process is called gene expression and different types of immune responses cause the activation of different genes.This study is looking at how specific parts of the immune system like B and T cells respond to the nasal spray vaccine and how and what genes are activated by the vaccine. B cells make antibodies, a part of our immune system that helps to protect against invaders such as viruses or bacteria. The next time our bodies are exposed to the same invader, our B cells make antibodies that can recognise and stop the invader going on to cause an infection. Our T cells can help B cells to make antibodies and also help to direct the body to attack the invader instead of causing harm to healthy cells.

DETAILED DESCRIPTION:
Influenza infection is related to significant morbidity and mortality in children. Although usually causing a self-limiting illness, the increased risk for children of hospitalisation and further complications, ranging from secondary pneumonia to death, reflect the need to focus on prevention. The commonly used trivalent inactive influenza vaccine (TIV) has been documented to have poor immunogenicity in children. The live attenuated influenza vaccine (LAIV) was introduced with the idea to induce superior protection than TIV. Early efficacy studies suggested that LAIV provides superior protection to TIV in children, however the mechanisms of action at a molecular and immunological level are not yet well described. This study aims to understand how the LAIV works from a gene expression and immunological perspective using a systems biology approach and relate these findings to adaptive immune responses and immunogenicity. Success of this study will yield the first comprehensive picture of cellular and molecular signature that underlie a successful response to LAIV vaccination in children.

The LAIV was introduced to provide broader protection by stimulation of both antibody and T cell responses. At present the two major obstacles in the widespread use of LAIV are concerns raised over its effectiveness and the lack of defined immunological correlates of protection. In this study, by identifying key genes and immune cells that are participating in the vaccine-induced responses, the investigators aim to understand molecular and immunological mechanism of LAIV.

In 2016 the Centers for Disease Control and Prevention in the Unites States (US) recommended against the use of LAIV due to its poor effectiveness in their analysis of the 2015/2016 season. However, the same vaccine, in the same season had high effectiveness as assessed by two public health authorities in UK and Finland. Currently the reason for this discrepancy is not known. The annual childhood influenza vaccine programme in UK started in the 2013/2014 influenza season by the introduction of the newly licensed LAIV. Eligible healthy children were offered a single dose of LAIV, while children in a clinical risk group up to 9 years of age were offered two doses of vaccine. By the 2016/2017 season, the LAIV became a licensed vaccine in the UK for children and adolescents from 2 to 18 years of age. The UK has found evidence of LAIV effectiveness in 2015/2016 season of 58% and therefore it continues to recommend its use.

In this study, the investigators will administer LAIV to cohorts of children and investigate the immunological basis for the observed variability and define the role of adaptive immunity by applying the systems biology tools and machine learning algorithms for predictive modelling. Tracing the influenza vaccine imprint on immune system, termed FluPRINT, by the proposed project will help to identify cellular signatures of vaccine-induced protection in young children, which is of critical importance for the development of a new generation of influenza vaccines that will be more effective in this target population.

This project will cover an issue that has been poorly studied in humans and that is the role of influenza-specific T cells after vaccination. Correlating the cellular signature and T cell repertoire after vaccination with the vaccine efficacy is a novel approach to the current problem about usage of LAIV. Results obtained are expected to increase the understanding of the mechanisms of influenza vaccine effectiveness, by exploring for the first time the impact of vaccines on the influenza-specific T cell repertoire in children while their adaptive immune system is still being developed.

Despite many years on the market, no correlates of protection for LAIV have been defined. Recent studies using systems biology and computational methods identified baseline frequency of B and T cells to predict antibody responses on day 28 after TIV vaccination. A similar approach to define cellular signatures driving immunity to LAIV has not yet been reported. The current study aims to assess the detailed phenotypical and functional analysis of immune cells (focusing on T and B cells) combined with the molecular signature which will provide insights into LAIV's mechanisms of protection. To comprehensively probe the phenotypic and functional profiles of different immune cells, in the proposed study the investigators will analyse blood samples in children aged 4-6 years before and 28 days after LAIV vaccination using mass cytometry (CyTOF), Luminex and transcriptome analysis which will be correlated with HAI titers. This study will be an exploratory study with between 30 and 40 children allocated to 4 groups; Group 1: up to 10 children aged 4-6 years that never received LAIV before. Group 2: up to 10 children aged 4-6 years that received LAIV once before, Group 3: up to 10 children aged 4-6 years that were vaccinated twice before and Group 4: up to 10 children aged 4-6 years vaccinated 3 or 4 times.

ELIGIBILITY:
Inclusion Criteria:

* The investigator believes that the parents/LAR(s) of the child can and will comply with requirements of the protocol (e.g. understanding of study procedure, consent process, availability at visits).
* Written informed consent obtained from parent(s)/LAR(s) of the subject
* Age from 4y+ 1day up to 6 years (until the day they turn 7y) at time of V1 (first immunisation visit)
* Born to two white Caucasian (of European descent) parents
* Participant is healthy as determined by general health assessment
* Have received all the vaccines specified in the UK immunisation schedule
* Group 1: Never received the intranasal flu vaccine before
* Group 2: Must have had at least 1 dose of the intranasal flu vaccine
* Group 3: Must have had at least 2 doses of the intranasal flu vaccine
* Group 4 : Must have had at least 3 or 4 doses of the internasal flu vaccine

Exclusion Criteria:

* Use (or planned use) of any non-registered or investigational product in 30 days before or after study vaccination
* Chronic serious medical conditions which may, in the opinion of the investigator, interfere with evaluation of study objectives e.g. chronic lung disease, chronic liver/renal disease, chronic renal failure chronic heart disease, congenital genetic syndromes (e.g. Trisomy 21).
* Recommended for inactivated influenza vaccine in UK (e.g. Children in clinical risk groups as specified by Public Health England) according to the Green Book, DoH.
* Meets any contraindications to vaccination as outlined in the Green Book, DoH
* Suspected or confirmed immunosuppressive or immunodeficiency conditions (including splenic dysfunction & HIV)
* Autoimmune conditions (e.g. Type 1/2 diabetes mellitus, thyroid disease, juvenile idiopathic arthritis) and bleeding disorders
* Use of systemic steroids for more than one week e.g. prednisolone >0.5mg/kg/day in the three months prior to first study intervention
* Chronic administration (≥14 days in total) of immunosuppressant's or other immune modifying drugs in the 3 months prior to first study intervention
* Receipt of blood, blood products and/or plasma derivatives or any immunoglobulin preparation in the three months prior to first study intervention

Temporary exclusion criteria:

* Participants who have experienced fever (≥38.0°C) or coryzal symptoms within the 24 hours prior to first study intervention
* Actively wheezing or increased bronchodilators in the previous 72 hours prior to first study intervention
* Immunisation with inactivated vaccines within the week prior to first study intervention, or live vaccines within the three weeks prior to first study intervention
* Receipt of antipyretics within six hours prior to immunisation

Ages: 48 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
To assess the change in molecular signature from baseline to day 28 after LAIV vaccination | Baseline and day 28 after vaccination
  To assess gene expression differences between participants at baseline and day 28 after vaccination.
To assess the change in immunological signature from baseline to day 28 after LAIV vaccination | Baseline and day 28 after vaccination
  To assess differences in the phenotype and frequency of immune cell subsets analyzed by 40-antibody panel mass cytometry between participants at baseline and day 28 after vaccination.
To assess the change in HAI antibody titer from baseline to day 28 after LAIV vaccination | Baseline and day 28 after vaccination
  Percentage of participants with a 4 fold rise in HAI titre between the baseline sample and sample taken on day 28 after vaccination and percentage of participants with the HAI titer above 40.

SECONDARY OUTCOMES:
To assess the change in functionality of the adaptive immune responses to LAIV from baseline to day 28 after LAIV vaccination | Baseline and day 28 after vaccination
  To assess the differences in activation and intracellular cytokine secretion of CD4+, CD8+ T cells and B cells after influenza peptide library stimulation in PBMC samples before and on day 28 after vaccination between participants.
To analyze the change in the influenza-specific T-cell repertoire (TCR) from baseline to day 28 after LAIV vaccination | Baseline and day 28 after vaccination
  To assess the TCR repertoire changes between baseline and day 28 post-vaccination using single-cell sequencing of sorted influenza-specific T cells identified using activation markers (CD137 and CD154) after influenza peptide library stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, FRCPCH, Study Chair — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No